CLINICAL TRIAL: NCT01646450
Title: An Open Lable, Single Arm, Phase IV Study of Icotinib as First-line Treatment in Elder NSCLC Patients With EGFR Mutation
Brief Title: First-line Treatment With Icotinib in Elder NSCLC EGFR Mutated Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV20
Record Dates: First submitted 2012-07-17; First posted 2012-07-20 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: NSCLC; EGFR Mutation; Elder patients
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Icotinib (Experimental): Icotinib: 125mg, oral administration, three times per day.
  Interventions: Drug: Icotinib

INTERVENTIONS:
Drug: Icotinib — Icotinib: 125mg, oral administration, three times per day.
  Other Names: BPI-2009; Commana

SUMMARY:
A single arm, open label, phase IV trial to evaluate safety and efficacy of icotinib as first-line treatment for the elder patients with advanced or metastatic (IIIb and IV) NSCLC and mutated EGFR.

DETAILED DESCRIPTION:
A single arm, open label, prospective, phase IV trial to evaluate safety and efficacy of icotinib as first-line treatment for the elder patients with advanced or metastatic (IIIb and IV) NSCLC and mutated EGFR.

* Primary endpoint to assess progression-free survival
* Secondary endpoints to assess the overall survival, objective response rate, disease control rate and so on.

ELIGIBILITY:
Inclusion Criteria:

* Recurrent or progressive Non-Small Cell Lung Cancer stage IV or IIIB patients.
* Positive EGFR Mutation.
* No previous systemic anticancer therapy.
* Male and female patients aged over 70 years.
* Measurable lesion according to RECIST with at least one measurable lesion not previously irradiated, unless disease progression has been documented at that site.
* Provision of written informed consent.

Exclusion Criteria:

* Evidence of clinically active Interstitial Lung Diseases (Patients with chronic, stable, radiographic changes who are asymptomatic need not be excluded).
* Known severe hypersensitivity to icotinib or any of the excipients of this product.
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the study.

Ages: 70 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2012-07; Primary Completion 2015-12 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 12 months
  PFS was defined as the time from the date of first dose of study medication to the date of first documentation of tumor progression or death due to any cause, whichever occurred first.

SECONDARY OUTCOMES:
Overall survival | 24 months
  Overall Survival was assessed via calculation of the time to death due to any cause. If a participant was known to have died, the time to death was defined as the time from the date of randomization to the date of death. Otherwise, a participant was censored at the last date they were known to be alive.
Objective response rate | 3-6 months
  Number of participants with an objective response. An objective response (OR) was defined as a patient having a best overall response of either complete response (CR) or partial response (PR) according to RECIST, confirmed at least 28 days following the date of the initial response.
Number of Participants with Adverse Events as a Measure of Safety | 18 months
  Adverse events, Serious adverse events , incidence of and reason for study drug dose interruptions and discontinuations, laboratory assessments, vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Han Baohui, MD, Principal Investigator — Shanghai Chest Hospital Affliated to Shanghai Jiaotong Univercity
Locations (1):
- Shanghai Chest Hospital Affliated to Shanghai Jiaotong Univercity, Shanghai, Shanghai Municipality, China